CLINICAL TRIAL: NCT06744660
Title: Clinical Validation of the Aptitude Medical Systems Metrix COVID-19 Test for Detection of SARS-CoV-2 in Point-of-Care and At-Home (OTC)/Non-Laboratory Settings
Brief Title: Clinical Validation of the Aptitude Medical Systems Metrix COVID-19 Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aptitude Medical Systems (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP-24-028
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; COVID
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OTC Study (Experimental): This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.
  Interventions: Diagnostic Test: Aptitude Medical Systems Metrix COVID Test

INTERVENTIONS:
Diagnostic Test: Aptitude Medical Systems Metrix COVID Test — The Metrix COVID Test is a real-time reverse transcription loop-mediated isothermal amplification reaction (RT-LAMP) test that has been designed to detect viral RNA from SARS-CoV-2 via electrochemical detection using the Metrix Reader. Detection of SARS-CoV-2 gene targets will produce a positive SARS-CoV-2 result. If no target is detected and the internal control amplifies, the result is negative. If no amplification is detected in any of the channels, an invalid result is displayed.

SUMMARY:
The Metrix COVID Test will be evaluated for use in Point-of-Care and Non-Laboratory settings in a home testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix COVID Test for the detection of SARS-CoV-2 AN swab samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for the detection of SARS-CoV-2.

DETAILED DESCRIPTION:
The Metrix COVID Test will be evaluated for OTC use in a home use testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix COVID Test for the differential detection of SARS-CoV-2 in AN swab samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for detection of SARS-CoV-2.

The candidate device, Metrix COVID Test, will be evaluated with AN swab sample types. Each Metrix COVID Test kit contains all supplies needed to test AN swab samples, including a corresponding QRI for detailed instructions.

This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.

For each participant, a comparator NP swab sample will be obtained by a healthcare practitioner after testing with the candidate device. This NP swab will be tested with the FDA-cleared SARS-CoV-2 assay according to the IFU and will serve as the primary comparator for swab samples. An additional AN swab sample will be collected and stored frozen and dry for later analysis to support future research validation studies.

No results from the investigational test or comparator testing will be used for clinical diagnosis, management of study participants, or to make treatment decisions.

Test results from the Metrix COVID Test (investigational test) will be compared to the test results generated from the comparator assay.

No investigational test results will be reported to a third party or used for any treatment decisions.

This work is supported by funding provided by the Biomedical Advanced Research and Development Authority (BARDA).

ELIGIBILITY:
Inclusion Criteria:

1. Participant or guardian understands and is able and willing to provide written informed consent, and assent where applicable, prior to study enrollment.
2. Male or female aged 2 years or older
3. Participant is currently exhibiting fever, or one or more symptoms of respiratory tract infection (such as, but not limited to, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting or diarrhea). Participant must still be exhibiting symptoms on the day of sample collection.
4. Participant or guardian agrees to read, and is able to read with understanding, the AN swab QRI prior to beginning the operation of each of the Metrix COVID-19 Test.
5. Participant or guardian is able and willing to contribute the required swab samples for testing and understands and is able and willing to sign the study informed consent.

Exclusion Criteria:

1. Participant does not understand and/or is not able and willing to sign the study informed consent and/or assent.
2. Participant or guardian is not able to comply with nasal swab collection requirements following the QRI.
3. Participant has previously provided a sample for the study.
4. Participant is not able to tolerate sample collection.
5. Participant is currently undergoing antiviral treatment such as baloxavir marboxil (trade name Xofluza®), oseltamivir (Tamiflu®), zanamivir (Relenza®), and peramivir (Rapivab®).
6. Participants currently undergoing treatment and/or within the past thirty (30) days with prescription medication to treat novel Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury), Paxlovid, molnupiravir or receiving convalescent plasma therapy for SARS-CoV-2.
7. Participants who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to the study sample collection.
8. Participants who have had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.
9. Participants who do not understand/read the English language.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative detection of RNA from SARS-CoV-2 and Measurement of Positive/Negative Percent Agreement with FDA-cleared comparator test | 25 minutes
  Qualitative detection of RNA from SARS-CoV-2 in unprocessed AN swab samples. Primary objective of this study is to evaluate the performance (positive percent agreement, negative percent agreement and 95% confidence intervals for upper and lower bounds) of the Metrix COVID/Flu Test for the qualitative detection of SARS-CoV-2 viral RNA using AN swab samples. Comparator testing will be performed to determine the status of each sample for comparison to results produced by the candidate test. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay that detects SARS-CoV-2.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AFC Montclair, Birmingham, Alabama
  - AFC Madison, Madison, Alabama
  - PPU Mid City, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided